CLINICAL TRIAL: NCT07385612
Title: RESEARCH ON FACTORS OF RESISTANCE TO CHEMOTHERAPY AND INNOVATIVE THERAPIES IN MATURE B-CELL LYMPHOIDS
Acronym: REFRACT-LyMA
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0358
Record Dates: First submitted 2026-01-21; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: MATURE B-CELL LYMPHOIDS
Keywords: B-cell non-Hodgkin lymphoma; treatments resistance; tumor microenvironment; biocollection
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed or relapsed NHL-B patients (based on ongoing translational research studies): Clinical data collection and blood, bone marrow, lymphadenopathy as well as pleural fluid and ascites sampling at the time of inclusion (for diagnosis or relapse) and at each relapse/progression.

SUMMARY:
In order to promote translational research on the molecular pathways involved in resistance to treatments for mantle cell lymphoma (MCL), the clinical haematology department of the University Hospital Center (CHU) of Nantes has established, since 2016, the REFRACT-LyMa (Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mantle Cell Lymphoma) cohort-biocollection of blood and bone marrow samples from patients with MCL. Thanks to the close collaborations with team 11 of the Integrated Cancer Research and Immunology Center Nantes Angers (CRCI²NA), which specializes in studying the molecular pathways involved in resistance to treatments for hematological cancers, we wish to broaden the scope of research to other B-cell non-Hodgkin lymphomas (B-NHL). That is why today the REFRACT-LyMa cohort-biocollection aims to expand to malignant hematopathies involving mature B cells (Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mature B-Cell Lymphoid Hemopathies).

DETAILED DESCRIPTION:
A collection of tumor samples collected before the initiation of any new line of treatment as well as after any relapse/progression, is essential to identify the factors of response or resistance to a given therapy. To support the translational research projects on MCL in collaboration with team 11 of CRCI²NA, the clinical hematology department of the CHU of Nantes established, in 2016, the prospective multicentric (five centers: Nantes, La Roche-sur-Yon, Vannes, Saint-Nazaire and Poitiers) cohort-biocollection REFRACT-LyMA (Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mantle Cell Lymphoma), with the aim of constituting a cohort of patients integrating clinico-biological data linked to a biocollection of blood, bone marrow, lymphadenopathy, pleural fluid and ascites samples. Thanks to primary cells from patients derived from the biocollection, the REFRACT-LyMa cohort has highlighted molecular aberrations and genomic instability of tumor cells leading to the emergence of heterogeneous subclones at the base of the main mechanism of chemoresistance, which can be used as predictive factors of response/sensitivity to treatments in MCL. However, the therapies used in MCL are also applicable to other malignant hematopathies. That is why we wish to expand our cohort-biocollection to the Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mature B-Cell Lymphoid Hemopathies (REFRACT-LyMa). Although the patients with MCL already included in the cohort "Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mantle Cell Lymphoma" will continue to be followed retrospectively and new MCL patients will be included prospectively, not all new patients with B-NHL will be automatically included in the new cohort "Research on Factors of Resistance to Chemotherapies and Innovative Therapies in Mature B Lymphoid Hemopathies". The choice will depend on the pathology subject to the ongoing translational research studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient affected by B-NHL (at diagnosis or relapse).
* Patient who has signed the consent form.
* Patient affiliated with a social security system.

Exclusion Criteria:

* Minor patients.
* Adults under guardianship.
* Protected persons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed or relapsed B-NHL patients managed in the hematology departments of Nantes, La Roche-Sur-Yon, Saint-Nazaire and Poitiers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Characterization of the tumor | 10 years
  Characterization of the tumor and its microenvironment in B-NHL in order to develop preclinical models of ex vivo culture and genetic modifications of primary B-NHL cells.

SECONDARY OUTCOMES:
Preclinical model | 10 years
  Development of preclinical models of ex vivo culture to analyze the response to treatment
Preclinical model | 10 years
  Development of genetic modifications of primary B-NHL cells to evaluate resistance mechanisms
Data analysis | 10 years
  Analysis of genomic data to identify resistance genes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No